CLINICAL TRIAL: NCT05983809
Title: Technological Balance and Gait Rehabilitation in Patients With Multiple Sclerosis: Effects on Functional, Motor and Cognitive Outcomes (ROAR-MS).
Brief Title: Technological Balance and Gait Rehabilitation in Patients With Multiple Sclerosis.
Acronym: ROAR-MS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, GIOVANNINI SILVIA, Principal investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 0000051/23
Record Dates: First submitted 2023-08-01; First posted 2023-08-09 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2024-12

CONDITIONS: Multiple Sclerosis; Balance; Cognitive Impairment
Keywords: Rehabilitation; Multiple Sclerosis; Technology; Balance; Cognitive Impairment
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Interventional, randomised, controlled, cross-over pilot study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (HO, Hunova-Observation) (Experimental): Patients in the HO group will undergo a specific rehabilitation treatment for balance disorders using the robotic platform Hunova® Movendo Technology srl, Genova, IT), for 4 weeks, 3 times a week for 45 minutes each. In particular, the technological rehabilitation carried out with the platform will have as main objective the improvement of balance, both in sitting and standing position, and static and dynamic exercises, dual-task exercises and exercises to improve trunk control will be proposed. Afterwards, patients will undergo 4 weeks of observation without rehabilitation treatment.
  Interventions: Device: Technological rehabilitation
- Control Group (OH, Observation-Hunova) (Active Comparator): Patients in the OH group will undergo 4 weeks of observation without rehabilitation treatment, followed by specific rehabilitation treatment for balance disorders using the robotic platform Hunova® Movendo Technology srl, Genova, IT), for 4 weeks, 3 times a week for 45 minutes each. In particular, the technological rehabilitation carried out with the platform will have as main objective the improvement of balance, both in sitting and standing position, and static and dynamic exercises, dual-task exercises and exercises to improve trunk control will be proposed.
  Interventions: Device: Technological rehabilitation

INTERVENTIONS:
Device: Technological rehabilitation — Specific rehabilitation for balance disorder using the robotic platform
  Other Names: Hunova® MovendoTechnology srl

SUMMARY:
Multiple sclerosis (MS) is a chronic, inflammatory and neurodegenerative disease of the central nervous system that often results in motor and/or cognitive impairment. Epidemiologically, the onset occurs between the ages of 20 and 40, with a peak around the age of 30.

MS is an extremely heterogeneous disease in terms of signs and symptoms, both in terms of the neurological systems involved and the degree of impairment and severity. The most common symptoms include, among others, difficulty walking and lack of balance. The lack of stability and coordination reduces independence and mobility, predisposing people with MS to accidental falls and compromising mobility in daily life. Another symptom that characterises MS is cognitive impairment, which mainly alters information processing speed and short- and long-term memory. MS-related cognitive impairment is detectable at every stage of the disease. Very often, people with MS have co-existing cognitive and motor deficits, which add to the complexity of managing MS. In order to address this condition, a treatment strategy that combines cognitive and motor rehabilitation needs to be identified. Despite the increasing availability of effective drug therapies that may impact on balance, rehabilitation is a very important means to counteract the progression of disability and improve physical function, affecting social participation and improving quality of life. In recent years, rehabilitation makes use of various robotic devices, which are based on repeatable, intense and motivating exercises, integrated with an enriched virtual environment, capable of improving the quality of movement. In light of the literature, which mainly focuses on robotic therapy for walking, this pilot study aims to evaluate the effects of a specific robotic treatment for balance in MS patients.

The primary objective of the study is the evaluation of the effects of technological rehabilitation by means of a robotic platform (Hunova® Movendo Technology srl, Genoa, IT) on static balance.

The secondary objective is the evaluation of the effects of technological rehabilitation by means of a robotic platform (Hunova® Movendo Technology srl, Genoa, IT)

1. on dynamic balance and walking (assessed with clinical and instrumental scales)
2. on fatigue and cognitive performance in terms of sustained attention, dual-task cost and cognitive-motor interference;
3. on quality of life.

DETAILED DESCRIPTION:
Twenty-four patients of both sexes will be recruited, evaluated and treated at the Multiple Sclerosis UOS of the Fondazione Policlinico Universitario Agostino Gemelli IRCCS in Rome from the date of approval of the study by the ethics committee and for the following 12 months, meeting the inclusion criteria. Patients will be divided into two groups by randomisation: one group (experimental group, HO, Hunova-Observation) will perform specific rehabilitation for balance disorder using the robotic platform Hunova® Movendo Technology srl, Genova, IT), followed by 4 weeks of observation. The other group (OH, Observation-Hunova) will instead carry out 4 weeks of observation, at the end of which they will carry out the specific treatment for the balance disorder using the robotic platform Hunova® Movendo Technology srl, Genova, IT).

ELIGIBILITY:
Inclusion Criteria:

* Definitive diagnosis of multiple sclerosis according to McDonald criteria;
* Age between 18 and 65 years;
* Pyramidal or cerebellar system with a score ≥ 2 on the EDSS;
* EDSS between 2 and 3;
* Ability to stand without support for 60 seconds;
* Stability of disease-modifying treatment and absence of clinical relapse of the disease for at least 1 year;
* Cognitive ability to execute simple orders and understand the physiotherapist's instructions [assessed by Token Test (score ≥ 26.5)];
* Ability to understand and sign informed consent.

Exclusion Criteria:

* Significant visual impairment, defined by a visual system score ≥ 2 on the EDSS;
* Presence of vestibular disorders unrelated to MS;
* Presence of psychiatric disorders or severe cognitive impairment, i.e. a Mini Mental State Examination (MMSE) score < 24 (15);
* Presence of cardiovascular and respiratory disorders;
* Inability to provide informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale | Change from Baseline BBS at 4 and 8 weeks
  The Berg Balance Scale (BBS) is used to objectively determine a patient's ability(or inability) to safely balance during a series of predetermined tasks. It is a 14item list with each item consisting of a five-point ordinal scale ranging from 0 to 4,with 0 indicating the lowest level of function and 4 the highest level of function andtakes approximately 20 minutes to complete. It does not include the assessmentof gait.

SECONDARY OUTCOMES:
Modified Fatigue Impact Scale (MFIS) | Change from Baseline MFIS at 4 and 8 weeks
  The Modified Fatigue Impact Scale (MFIS) is an instrument that provides anassessment of the effects of fatigue in terms of physical, cognitive, andpsychosocial functioning. The full-length MFIS consists of 21 items while theabbreviated version has 5 items.
  The MFIS is a structured, self-report questionnaire that the patient can generallycomplete with little or no intervention from an interviewer. However, patients withvisual or upper extremity impairments may need to have the MFIS administeredas an interview. Interviewers should be trained in basic interviewing skills and inthe use of this instrument.
  The total score for the MFIS is the sum of the scores for the 21 items. Individualsubscale scores for physical, cognitive, and psychosocial functioning can also begenerated by calculating the sum of specific sets of items.
Fatigue Scale for Motor and Cognitive Function (FSMC) | Change from Baseline FSMC at 4 and 8 weeks
  The FSMC is an assessment of MS-related cognitive and motor fatigue. A Likert-type 5-point scale (ranging from 'does not apply at all' to 'applies completely')produces a score between 1 and 5 for each scored question. Thus minimumvalue is 20 (no fatigue at all) and maximum value is 100 (severest grade offatigue). Two subscales (mental and physical fatigue) can be made. Items included in the subscale mental are 1-4-7-8-11-13-15-17-18-20 and items included in the subscale physical are 2-3-5-6-9-10-12-14-16-19.
Timed Up and Go test (TUG) | Change from Baseline TUG at 4 and 8 weeks
  The Timed Up and Go test (TUG) measures in seconds the time it takes a subjectto rise from a chair, walk a distance of 3 meters, turn, walk back to the chair andsit down.
  The performance is rated on a scale of 1 to 5 (where 1 is normal and 5 is severelyabnormal) according to the observer's perception of the patient's risk of falling.
  The timed part of the test records the mean time (in seconds) from initial gettingup to re-seating. Patients are compared with the mean time of adults in their agegroup, 60 to 69, 70 to 79, and 80 to 99 years of age.
Ambulation Index (AI) | Change from Baseline Ambulation Index at 4 and 8 weeks
  Ambulation Index (AI) The Ambulation Index is a rating scale to assess mobility by evaluating the timeand degree of assistance required to walk 8 meters. Scores range from 0(asymptomatic and fully active) to 10 (bedridden). The patient is asked to walk amarked 8 meters course as quickly and safely as possible. The examiner recordsthe time and type of assistance (e.g., cane, walker, crutches) needed. Althoughthe patient's walking is timed, the time is not used directly but is utilized inconjunction with other factors to rate the patient on an ordinal scale with 11gradations.
  0 = Asymptomatic; fully active. 10 = Bedridden
Walking handicap scale (WHS) | Change from Baseline Walking handicap scale at 4 and 8 weeks
  The Walking handicap scale (WHS) is an assessment tool that allows us toevaluate the quality of walking in the home and social environment through a ascale comprising six categories.
  1 = Physiological walking: walking only as exercise 6 = Unrestricted walking insocial settings: independent in all activities, on uneven ground, in crowded places,shows complete independence in public places
Functional Ambulation Classification (FAC) | Change from Baseline Functional Ambulation Classification at 4 and 8 weeks
  The Functional Ambulation Categories (FAC) is a functional walking test thatevaluates ambulation ability. This 6-point scale assesses ambulation status bydetermining how much human support the patient requires when walking,regardless of whether or not they use a personal assistive device.
  A score of 0 indicates that the patient is a non-functional ambulator (cannot walk);A score of 1, 2 or 3 denotes a dependent ambulator who requires assistance fromanother person in the form of continuous manual contact (1), continuous orintermittent manual contact (2), or verbal supervision/guarding (3).
  A score of 4 or 5 describes an independent ambulator who can walk freely on:level surfaces only (4) or any surface (5=maximum score).
10 Meter Walk Test (10mWT) | Change from Baseline 10 Meter Walk Test at 4 and 8 weeks
  The 10mWT is used to assess walking speed in meters/second (m/s) over a shortdistance. The total time taken to ambulate 6 meters (m) is recorded to the nearesthundredth of a second. 6 m is then divided by the total time (in seconds) taken toambulate and recorded in m/s.
  The time is measured for the middle 6 m to allow for patient acceleration anddeceleration.
  The time is started when any part of the leading foot crosses the plane of the 2-mmark.
  The time is stopped when any part of the leading foot crosses the plane of the 8-m mark.1 The time to walk the middle 6m, the level of assistance, and type ofassistive device and/or bracing used will be documented.
  If a patient requires total assistance or is unable to ambulate at all, a score of 0m/s will be documented.
Six-minute walk test (6MWT) | Change from Baseline Six-minute walk test at 4 and 8 weeks
  The six-minute walk test (6MWT) is a sub-maximal exercise test used to assesswalking endurance and aerobic capacity. Participants will walk around theperimeter of a set circuit for a total of six minutes. The score of the test is thedistance a patient walks in 6 minutes (measured in meters and can round to thenearest decimal point).
  Distance (in meters) covered in six minutes is calculated by multiplying thenumber of total laps by 12 meters and adding the distance of the partial lapcompleted at the time the test ended.
Multiple Sclerosis Walking Scale (MSWS-12) | Change from Baseline Multiple Sclerosis Walking Scale at 4 and 8 weeks
  The Multiple Sclerosis Walking Scale (MSWS-12) is a self-reported 12-item measure of an individual's ability to walk.
  Each item can be assigned a score from 1 to 5, where 1 means "no limitation" and 5 means "extreme limitation".
  The total score is obtained by summing the scores of the individual items; higher scores indicate a greater impact on walking than lower scores.
Modified Barthel Index (mBI) | Change from Baseline mBI at 4 and 8 weeks
  The modified Barthel Index (mBI) for activities of daily living is meant to be used in theassessment of patient performance (or degree of assistance required) with respect toself-care, sphincter management, transfers and locomotion. The index consist of 10items (each scored with a number of points) that relate to activities of daily living (ADLs)where the final score is calculated by summing the points awarded to each item. A five-point rating scales for each item to improve sensitivity to detecting change.
  The 10 items assessed relate to help needed with feeding, bathing, grooming, dressing,transfers, walking, climbing stairs, presence or absence of fecal incontinence and urinaryincontinence.
  The score ranges from 0 (maximum dependence) to 100 (maximum independence)
Multiple Sclerosis Impact Scale (MSIS-29) | Change from Baseline MSIS-29 at 4 and 8 weeks
  The 29-item Multiple Sclerosis Impact Scale (MSIS-29) is a self-administered questionnaire consisting of 20 physical and 9 psychological items to assess the impact of the disease on activities of daily living.
  For each item, it is possible to assign a score ranging from 1, "Not at all", to a maximum of 5, "Extremely".
  The total score is obtained by summing the scores for each item and can range from a minimum of 29, the minor impact of MS, to a maximum of 145, the extreme impact of MS.
Beck Depression Inventory-II (BDI-II) | Change from Baseline BDI-II at 4 and 8 weeks
  The Beck Depression Inventory-II (BDI-II) is a scale consisting of 21 items identified in four increasing levels of severity, and is specifically designed to measure the 'behavioural manifestations of depression'. The quantification criteria are well defined for each item, and in fact, each severity level corresponds to a specific definition from which patients had to choose the one that best described their situation, taking into account the period including the last week before the test. At the end of the compilation, summing up the scores of the 21 items, which range from 0 to 3, gives four different degrees of depression:
  * Scores between 0 and 10 indicate the absence of depressive content;
  * Scores between 11 and 18 indicate mild depression;
  * Scores between 19 and 29 indicate moderate depression;
  * Scores between 30 and 63 indicate severe depression.
State-Trait Anxiety Inventory (STAI-Y1 and Y2) | Change from Baseline STAI-Y1 and Y2 at 4 and 8 weeks
  The State-Trait Anxiety Inventory (STAI-Y) is a scale used to assess state and trait anxiety. The STAI-Y is subdivided into two scales (Y1 and Y2), which respectively assess state anxiety, with questions that relate to how the subject feels at the time the questionnaire is administered, and trait anxiety, with questions that investigate how the subject habitually feels.
  The STAI-Y consists of 40 items, 20 relating to state anxiety and 20 to trait anxiety. The patient's self-assessment is expressed in frequency using a Likert scale ranging from 0 to 4 points, where higher scores are positively correlated with higher levels of anxiety, while low scores indicate a mild form of anxiety.
  The total score is between 20 and 80, with a threshold value predictive of anxiety symptoms of 40. Specifically, there are severity criteria: 40 to 50 mild form, 50 to 60 moderate, greater than 60 severe.
Stroop Colour Word Test (SCWT) | Change from Baseline SCWT at 4 and 8 weeks
  The Stroop Color and Word Test (SCWT) is a neuropsychological test extensively usedto assess the ability to inhibit cognitive interference that occurs when the processing of aspecific stimulus feature impedes the simultaneous processing of a second stimulusattribute, well-known as the Stroop Effect. The subject is asked to read the words in thefirst task, to name colors in the second and third tasks. It is necessary to mark both anymistakes made but also the time spent on each task. The cut-off for the error interferenceeffect is 4.24, while the cut-off for the time interference effect is 36.92.
Symbol Digit Modalities Test (SDMT) | Change from Baseline SDMT at 4 and 8 weeks
  The Symbol Digit Modalities Test (SDMT) is a test that assesses information processing speed and consists of a series of nine printed symbols to which nine numbers correspond. After a 'training' phase, patients are asked to match as many symbols as possible to the corresponding number in just 90 seconds. As the test persons can give written or oral answers, the test is suitable for people with motor disabilities or speech disorders.
  The score is calculated by adding up the number of correct substitutions in the 90-second interval (maximum = 110). Interpretation results from normalising the categories of gender, age and education.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Giovannini, MD, phD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kamm CP, Uitdehaag BM, Polman CH. Multiple sclerosis: current knowledge and future outlook. Eur Neurol. 2014;72(3-4):132-41. doi: 10.1159/000360528. Epub 2014 Jul 30. PMID 25095894
- [Background] Martin CL, Phillips BA, Kilpatrick TJ, Butzkueven H, Tubridy N, McDonald E, Galea MP. Gait and balance impairment in early multiple sclerosis in the absence of clinical disability. Mult Scler. 2006 Oct;12(5):620-8. doi: 10.1177/1352458506070658. PMID 17086909
- [Background] Morris ME, Cantwell C, Vowels L, Dodd K. Changes in gait and fatigue from morning to afternoon in people with multiple sclerosis. J Neurol Neurosurg Psychiatry. 2002 Mar;72(3):361-5. doi: 10.1136/jnnp.72.3.361. PMID 11861697
- [Background] Cattaneo D, Jonsdottir J. Sensory impairments in quiet standing in subjects with multiple sclerosis. Mult Scler. 2009 Jan;15(1):59-67. doi: 10.1177/1352458508096874. Epub 2008 Oct 9. PMID 18845654
- [Background] Sosnoff JJ, Shin S, Motl RW. Multiple sclerosis and postural control: the role of spasticity. Arch Phys Med Rehabil. 2010 Jan;91(1):93-9. doi: 10.1016/j.apmr.2009.09.013. PMID 20103402
- [Background] Prosperini L, Castelli L. Spotlight on postural control in patients with multiple sclerosis. Degener Neurol Neuromuscul Dis. 2018 Apr 3;8:25-34. doi: 10.2147/DNND.S135755. eCollection 2018. PMID 30050386
- [Background] van Asch, P. Impact of mobility impairment in multiple sclerosis 2-patients' perspectives. European Neurological Review. 2011; 6(2), 115-120. https://doi.org/10.17925/ENR.2011.06.02.115
- [Background] Benedict RH, Cookfair D, Gavett R, Gunther M, Munschauer F, Garg N, Weinstock-Guttman B. Validity of the minimal assessment of cognitive function in multiple sclerosis (MACFIMS). J Int Neuropsychol Soc. 2006 Jul;12(4):549-58. doi: 10.1017/s1355617706060723. PMID 16981607
- [Background] Amato MP, Hakiki B, Goretti B, Rossi F, Stromillo ML, Giorgio A, Roscio M, Ghezzi A, Guidi L, Bartolozzi ML, Portaccio E, De Stefano N; Italian RIS/MS Study Group. Association of MRI metrics and cognitive impairment in radiologically isolated syndromes. Neurology. 2012 Jan 31;78(5):309-14. doi: 10.1212/WNL.0b013e31824528c9. Epub 2012 Jan 18. PMID 22262744
- [Background] Langdon DW. Cognition in multiple sclerosis. Curr Opin Neurol. 2011 Jun;24(3):244-9. doi: 10.1097/WCO.0b013e328346a43b. PMID 21519256
- [Background] Prosperini L, Tomassini V, Castelli L, Tacchino A, Brichetto G, Cattaneo D, Solaro CM. Exergames for balance dysfunction in neurological disability: a meta-analysis with meta-regression. J Neurol. 2021 Sep;268(9):3223-3237. doi: 10.1007/s00415-020-09918-w. Epub 2020 May 23. PMID 32447551
- [Background] Castelli L, Prosperini L, Pozzilli C. Balance worsening associated with nabiximols in multiple sclerosis. Mult Scler. 2019 Jan;25(1):113-117. doi: 10.1177/1352458518765649. Epub 2018 Mar 13. PMID 29533137
- [Background] Bowman T, Gervasoni E, Amico AP, Antenucci R, Benanti P, Boldrini P, Bonaiuti D, Burini A, Castelli E, Draicchio F, Falabella V, Galeri S, Gimigliano F, Grigioni M, Mazzon S, Mazzoleni S, Mestanza Mattos FG, Molteni F, Morone G, Petrarca M, Picelli A, Posteraro F, Senatore M, Turchetti G, Crea S, Cattaneo D, Carrozza MC; "CICERONE" Italian Consensus Group for Robotic Rehabilitation. What is the impact of robotic rehabilitation on balance and gait outcomes in people with multiple sclerosis? A systematic review of randomized control trials. Eur J Phys Rehabil Med. 2021 Apr;57(2):246-253. doi: 10.23736/S1973-9087.21.06692-2. Epub 2021 Feb 4. PMID 33541044
- [Background] Thompson AJ, Banwell BL, Barkhof F, Carroll WM, Coetzee T, Comi G, Correale J, Fazekas F, Filippi M, Freedman MS, Fujihara K, Galetta SL, Hartung HP, Kappos L, Lublin FD, Marrie RA, Miller AE, Miller DH, Montalban X, Mowry EM, Sorensen PS, Tintore M, Traboulsee AL, Trojano M, Uitdehaag BMJ, Vukusic S, Waubant E, Weinshenker BG, Reingold SC, Cohen JA. Diagnosis of multiple sclerosis: 2017 revisions of the McDonald criteria. Lancet Neurol. 2018 Feb;17(2):162-173. doi: 10.1016/S1474-4422(17)30470-2. Epub 2017 Dec 21. PMID 29275977
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Julious, S.A. 'Sample size of 12 per group rule of thumb for a pilot study'. Pharmaceutical Statistics. 2005. Vol 4. Pages 287-291.
- [Background] Mun EY, von Eye A, White HR. An SEM Approach for the Evaluation of Intervention Effects Using Pre-Post-Post Designs. Struct Equ Modeling. 2009 Apr 1;16(2):315-337. doi: 10.1080/10705510902751358. PMID 20228953
- [Background] MacCallum, R. C., Browne, M. W., & Sugawara, H. M. (1996). Power Analysis and Determination of Sample Size for Covariance Structure Modeling. Psychological Methods, 1, 130-149. https://doi.org/10.1037/1082-989X.1.2.130
- [Background] Hu LT, Bentler PM (1998). Fit indices in covariance structure modeling: Sensitivity to underparameterized model misspecification. Psychological Methods, 3(4), 424-453. doi: 10.1037/1082-989X.3.4.424
- [Background] Hu LT, Bentler PM (1999). Cutoff Criteria for Fit Indexes in Covariance Structure Analysis: Conventional Criteria versus New Alternatives. Structural Equation Modeling, 6, 1-55. doi: 10.1080/10705519909540118
- [Background] Burnham, K. P., and Anderson, D. R. (2004).Multimodel inference: understanding AIC and BIC in model selection. Sociol. Methods Res. 33, 261-304. doi: 10.1177/0049124104268644
- [Background] R Core Team (2021). R: A language and environment for statistical computing. R Foundation for Statistical Computing, Vienna, Austria. URL https://www.R-project.org/.
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660